CLINICAL TRIAL: NCT03961802
Title: Early and Systematic Shoulder Rehabilitation Following Cervical Lymph Node Dissection
Acronym: RESYSTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC17_0489
Record Dates: First submitted 2019-03-08; First posted 2019-05-23 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Rehabilitation
Keywords: Rehabilitation; shoulder dysfunction; cervical lymph node dissection; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systematic early rehabilitation (Experimental): systematic early rehabilitation
  Interventions: Other: sessions of shoulder rehabilitation
- without systematic rehabilitation (No Intervention): without systematic rehabilitation

INTERVENTIONS:
Other: sessions of shoulder rehabilitation — 3 sessions of shoulder rehabilitation per week for 3 months (36 sessions)
  Arms: systematic early rehabilitation

SUMMARY:
A prospective, monocentric, controlled, randomized study of systematic early shoulder rehabilitation following cervical lymph node dissection for the prevention and treatment of shoulder dysfunction.

DETAILED DESCRIPTION:
Pre-inclusion: information, collection of consent, collection of antecedents and biometric data, clinical examination (goniometric measurement and visual analogic scale of pain), collection of DASH, EORTC QLQ-C30 and H&N35 questionnaires.

Surgical intervention (J0) and randomization into 2 groups:

Group 1 - systematic early rehabilitation Group 2 - without systematic rehabilitation

M3, M6, M12: collection of complications, adjuvant treatments, number of physiotherapy sessions performed, clinical examination (goniometric measurement and visual analogic scale of pain), collection of DASH, EORTC QLQ- C30 and H&N35 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in the oral and written French language
* unilateral or bilateral cervical lymph node dissection preserving the accessory spinal nerve
* Karnofsky index ≥ 80%
* Age ≥ 18 years

Exclusion Criteria:

* cognitive disorders
* predictable difficulties in compliance with treatment and/or follow-up
* pre-existing pathology involving shoulder and its mobility, independent of head and neck cancer
* comorbidity preventing rehabilitation of the shoulder
* time to start rehabilitation after 6 weeks postoperatively
* pregnant women
* minors
* majors under guardianship
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Disabilities of Shoulder, Arm and Hand Questionnaire (DASH) | 6 months postoperatively (M6)
  The total score is reported. The score is between 0 and 100. The higher the score, the higher the disability.

SECONDARY OUTCOMES:
Disabilities of Shoulder, Arm and Hand Questionnaire (DASH) | 3 and 12 months postoperatively (M3 and M12)
  The total score is reported. The score is between 0 and 100. The higher the score, the higher the disability.
visual analog score for pain (M3, M6 and M12) | 3, 6 and 12 months postoperatively (M3, M6 and M12)
  The reported score is between 0 and 10. The higher the score, the higher the pain.
goniometric measurement of flexion and abduction of the shoulder | 3, 6 and 12 months postoperatively (M3, M6 and M12)
  Goniometric measurement will be performed using a Rippstein's Plurimeter, with standardized position and movement for each measurement:
  * Sitting on a chair, the bust is straight, arm hanging down the body.
  * The plurimeter is placed on the distal part of the arm.
  * The flexion is in the sagittal plane around a transverse axis in the frontal plane.
  * The abduction is in the frontal plane around an anteroposterior axis contained in the sagittal plane.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 3, 6 and 12 months postoperatively (M3, M6 and M12)
  EORTC QLQ-C30 questionnaire has 30 questions and includes the following scale:
  - health and overall quality of life, scale have a score between 0 and 100. A high score indicates the preservation of a good quality of life.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 3, 6 and 12 months postoperatively (M3, M6 and M12)
  EORTC QLQ-C30 questionnaire has 30 questions and includes the following scale:
  - operating scale, scale have a score between 0 and 100. A high score for this scale indicates the preservation of a good quality of life.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 3, 6 and 12 months postoperatively (M3, M6 and M12)
  EORTC QLQ-C30 questionnaire has 30 questions and includes the following scale:
  - scale of generic symptoms. scale have a score between 0 and 100. A high score for this scale indicates the presence of symptoms acting as factors of deterioration of certain aspects of the quality of life.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck cancer module (H&N35) | 3, 6 and 12 months postoperatively (M3, M6 and M12)
  EORTC QLQ-H&N35 questionnaire evaluates the specific symptoms of patients with head and neck cancers. It consists of 35 items including 7 subscales .
  subscale scores are reported, All items and scales give a score between 0 and 100.
  For each subscale, a high score indicates the presence of a large number of specific symptoms, acting as factors of deterioration of certain aspects of the quality of life.
evaluate the compliance of patients to rehabilitation | 12 months postoperatively (M12)
  (% of rehabilitation sessions performed over 36 sessions)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France